CLINICAL TRIAL: NCT02377921
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Sialic Acid Extended-Release Tablets in Patients With GNE Myopathy (GNEM) or Hereditary Inclusion Body Myopathy (HIBM)
Brief Title: Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Sialic Acid in Patients With Glucosamine (UDP-N-acetyl)-2-epimerase Myopathy (GNEM) or Hereditary Inclusion Body Myopathy (HIBM)
Acronym: GNEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX001-CL301
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Hereditary Inclusion Body Myopathy; Distal Myopathy With Rimmed Vacuoles; Distal Myopathy, Nonaka Type; GNE Myopathy
Keywords: GNE Myopathy; GNEM; HIBM; Nonaka; Hereditary Inclusion Body Myopathy; DMRV
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aceneuramic Acid Extended-Release (Ace-ER) (Experimental): Ace-ER 6 g/day, divided 3 times per day (TID) for 48 weeks.
  Interventions: Drug: aceneuramic acid extended-release (Ace-ER)
- Placebo (Placebo Comparator): Matching placebo TID for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aceneuramic acid extended-release (Ace-ER) — tablets for oral use
  Other Names: UX001; sialic acid extended-release (SA-ER)
  Arms: Aceneuramic Acid Extended-Release (Ace-ER)
Drug: Placebo — tablets for oral use
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of 6 g/day aceneuramic acid extended-release (Ace-ER) treatment of participants with GNEM on upper extremity muscle strength (upper extremity composite [UEC] score) as measured by dynamometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 55 years, inclusive
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and before any research-related procedures are conducted
* Have a documented diagnosis of GNEM, HIBM, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease due to previously demonstrated mutations in the gene encoding the GNE/N-acetylmannosamine kinase (MNK) enzyme (genotyping will not be conducted in this study)
* Able to provide reproducible force in elbow flexors (i.e. two dynamometry force values with no more than 15% variability in the dominant arm) at Screening
* Able to walk a minimum of 200 meters during the six-meter walk test (6MWT) at Screening without the use of assistive devices, including a cane, crutch(es), walker, wheelchair or scooter (ankle foot orthosis/orthoses are permitted)
* Willing and able to comply with all study procedures
* Participants of child-bearing potential or with partners of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use a highly effective method of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation, or true abstinence [when this is in line with the preferred and usual lifestyle of the subject], which means not having sex because the subject chooses not to), from the period following the signing of the informed consent through 3 months after last dose of study drug
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause for at least two years, have had tubal ligation at least one year prior to Screening, or who have had a total hysterectomy or bilateral salpingo-oophorectomy

Exclusion Criteria:

* Ingestion of N-acetyl-D-mannosamine (ManNAc), sialic acid (SA), or related metabolites; intravenous immunoglobulin (IVIG); or anything that can be metabolized to produce SA in the body within 60 days prior to the Screening Visit
* History of more than 30 days treatment with SA-ER and/or Sialic Acid Immediate Release (SA-IR) in prior clinical trials in the past year
* Has had any hypersensitivity to SA or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* Has serum transaminase (i.e. aspartate aminotransferase [AST] or gamma-glutamyl transpeptidase [GGT]) levels greater than 3X the upper limit of normal (ULN) for age/gender, or serum creatinine of greater than 2X ULN at Screening
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or anticipated requirement for any investigational agent prior to completion of all scheduled study assessments
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study
* Has a concurrent disease, active suicidal ideation, or other condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - University of California, Irvine, Irvine, California
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
- UMHAT "Alexandrovska", Sofia, Bulgaria
- McMaster University, Hamilton, Ontario, Canada
- France (2):
  - CHU La Réunion - site GHSR, Saint-Pierre, Reunion
  - Institut de Myologie GH Pitié-Salpêtrière, Paris
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- Italy (3):
  - University of Messina, Messina
  - University of Milan, Milan
  - Università Cattolica, Rome
- The Newcastle upon Tyne Hospitals, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Result] Lochmuller H, Behin A, Caraco Y, Lau H, Mirabella M, Tournev I, Tarnopolsky M, Pogoryelova O, Woods C, Lai A, Shah J, Koutsoukos T, Skrinar A, Mansbach H, Kakkis E, Mozaffar T. A phase 3 randomized study evaluating sialic acid extended-release for GNE myopathy. Neurology. 2019 Apr 30;92(18):e2109-e2117. doi: 10.1212/WNL.0000000000006932. Epub 2019 Jan 25. PMID 31036580
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971

RESULTS

PARTICIPANT FLOW:
Groups:
- Ace-ER 6 g/Day: Aceneuramic acid extended-release (Ace-ER) 6 g/day, divided 3 times per day (TID) for 48 weeks.
Period: Overall Study
Arm/Group | Ace-ER 6 g/Day | Placebo
Started | 45 | 44
Completed | 44 | 43
Not Completed | 1 | 1
Not completed — Subject non-compliance | 1 | 1

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement
Groups:
- Ace-ER 6 g/Day: Ace-ER 6 g/day, divided TID for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Ace-ER 6 g/Day | Placebo | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (7.91) | 36.2 (8.59) | 35.0 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 39 | 33 | 72
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 32 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Upper Extremity Composite (UEC) Score [Mean (Standard Deviation); unit: kg] — Muscle strength based on the maximum voluntary isometric contraction (MVIC) against a dynamometer was measured bilaterally in the following upper extremity muscle groups: gross grip, shoulder abductors, elbow flexors, and elbow extensors. The UEC is derived from the sum of the average of the right and left total force values (measured in kg).
  kg | 55.99 (26.950) | 56.31 (29.287) | 56.14 (27.954)
Muscle Strength in the Knee Extensors [Mean (Standard Deviation); unit: kg] — Lower extremity muscle strength in the knee extensors was measured by dynamometry. Bilateral total force was defined as the average of the right and left force values (measured in kg).
  kg | 26.53 (9.035) | 26.65 (8.969) | 26.59 (8.951)
Lower Extremity Composite (LEC) Score [Mean (Standard Deviation); unit: kg] — Muscle strength based on MVIC against a dynamometer was measured bilaterally in the following lower extremity muscle groups: knee flexors, hip flexors, hip extensors, hip abductors and hip adductors. The LEC is derived from the sum of the average of the right and left total force values (measured in kg).
  kg | 53.52 (33.751) | 55.17 (39.324) | 54.33 (36.378)
Glucosamine (UDP-N-acetyl)-2-epimerase Myopathy Functional Activities Scale(GNEM-FAS) Mobility Score [Mean (Standard Deviation); unit: units on a scale] — Lower extremity use and function was assessed using the Mobility domain of the GNEM-FAS instrument a disease specific measure developed to assess the functional impact of changes in muscle strength on mobility (reflective of the lower extremities). This mobility score ranges from 0 to 40 with higher scores representing greater mobility.
  units on a scale | 26.38 (7.581) | 26.23 (6.403) | 26.31 (6.990)
Stands in Sit-to-Stand Test [Mean (Standard Deviation); unit: stands] — Lower extremity function was assessed using a sit-to-stand test. The number of times the participant can rise from a seated to a standing position in a 30-second period was recorded.
  stands | 12.38 (4.103) | 12.58 (4.316) | 12.48 (4.185)
Lifts in Weighted Arm Lift Test [Mean (Standard Deviation); unit: arm lifts] — Upper extremity function was assessed using a weighted arm lift test performed bilaterally. The number of times the subject can raise a 1 kg weight above the head in a 30-second period was recorded.
  arm lifts | 30.50 (10.452) | 28.18 (9.824) | 29.33 (10.137)
Distance Walked in 6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — The total distance walked (meters) in a 6-minute period was measured.
  meters | 367.0 (115.07) | 361.2 (109.87) | 364.2 (111.95)
Percent of Predicted Distance Walked in 6MWT [Mean (Standard Deviation); unit: percentage of predicted meters] — The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated. Predicted Six-Minute Walk Test Distance (meters) = 868.8 - (2.99 x Age) - (74.7 x Sex), where Age is baseline age in years, and Sex = 0 for males, and 1 for females.
  percentage of predicted meters | 49.97 (15.521) | 49.87 (14.823) | 49.92 (15.097)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in UEC Score (Total Force in kg) at Week 48
Description: Muscle strength based on the maximum voluntary isometric contraction (MVIC) against a dynamometer was measured bilaterally in the following upper extremity muscle groups: gross grip, shoulder abductors, elbow flexors, and elbow extensors. The UEC is derived from the sum of the average of the right and left total force values (measured in kg).
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
kg | -2.25 [-3.77 to -0.74] | -2.99 [-4.69 to -1.28]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.5387, GEE model — Generalized estimating equation (GEE) model includes change from Baseline (BL) as dependent variable, visit, treatment and visit by treatment as fixed factors, and BL values, sex, and region as covariates, with compound symmetry covariance structure; Least Squares (LS) Mean Difference = 0.74, 95% CI 2-sided [-1.61 to 3.09] — Difference = Ace-ER - placebo

2. Secondary Outcome: Change From Baseline in Muscle Strength in the Knee Extensors at Week 48
Description: Lower extremity muscle strength in the knee extensors was measured by dynamometry. Bilateral total force was defined as the average of the right and left force values (measured in kg).
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
kg | 0.05 [-1.19 to 1.29] | 0.45 [-1.20 to 2.10]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.6938, GEE model — GEE model includes change from Baseline as dependent variable, visit, treatment and visit by treatment as fixed factors, and Baseline values, sex, and region as covariates, with compound symmetry covariance structure; LS Mean Difference = -0.40, 95% CI 2-sided [-2.38 to 1.58] — Difference = Ace-ER - placebo

3. Secondary Outcome: Change From Baseline in LEC Score (Total Force in kg) at Week 48
Description: Muscle strength based on MVIC against a dynamometer was measured bilaterally in the following lower extremity muscle groups: knee flexors, hip flexors, hip extensors, hip abductors and hip adductors. The LEC is derived from the sum of the average of the right and left total force values (measured in kg).
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
kg | -1.92 [-4.49 to 0.65] | -0.44 [-3.96 to 3.09]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.5023, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1.49, 95% CI 2-sided [-5.83 to 2.86] — Difference = Ace-ER - placebo

4. Secondary Outcome: Change From Baseline in GNEM FAS Mobility Domain Score at Week 48
Description: Lower extremity use and function was assessed using the Mobility domain of the GNEM-FAS instrument a disease-specific measure developed to assess the functional impact of changes in muscle strength on mobility (reflective of the lower extremities). This mobility score ranges from 0 to 40 with higher scores representing greater mobility.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
units on a scale | -2.49 [-3.56 to -1.42] | -1.77 [-2.59 to -0.95]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.2739, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.72, 95% CI 2-sided [-2.01 to 0.57] — Difference = Ace-ER - placebo

5. Secondary Outcome: Change From Baseline in Number of Lifts in the 30 Second Weighted Arm Lift Test at Week 48
Description: Upper extremity function was assessed using a weighted arm lift test performed bilaterally. The number of times the participant can raise a 1 kg weight above the head in a 30-second period was recorded.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: arm lifts
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
arm lifts | 0.03 [-2.19 to 2.26] | 2.79 [0.21 to 5.38]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.1235, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -2.76, 95% CI 2-sided [-6.27 to 0.75] — Difference: Ace-ER 6 g/day - placebo

6. Secondary Outcome: Change From Baseline in Number of Stands in the Sit to Stand Test at Week 48
Description: Lower extremity function was assessed using a sit-to-stand test. The number of times the participant can rise from a seated to a standing position in a 30-second period was recorded.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: stands
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
stands | 0.11 [-0.55 to 0.77] | 0.53 [-0.21 to 1.28]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.3907, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.43, 95% CI 2-sided [-1.40 to 0.55] — Difference: Ace-ER 6 g/day - placebo

7. Secondary Outcome: Change From Baseline in Meters Walked in the 6MWT at Week 48
Description: The total distance walked (meters) in a 6-minute period was measured.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
meters | -17.79 [-32.09 to -3.50] | -6.81 [-16.83 to 3.21]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Other; p = 0.1964, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -10.98, 95% CI 2-sided [-27.64 to 5.68] — Difference: Ace-ER 6 g/day - placebo

8. Secondary Outcome: Change From Baseline in Percent Predicted Meters Walked in the 6MWT at Week 48
Description: The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted meters
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
percentage of predicted meters | -2.37 [-4.30 to -0.44] | -0.97 [-2.32 to 0.38]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Superiority; p = 0.2241, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1.40, 95% CI 2-sided [-3.66 to 0.86] — Difference: Ace-ER - placebo

9. Secondary Outcome: Change From Baseline in GNEM FAS Upper Extremity Domain Score at Week 48
Description: Upper extremity use and function was assessed using the Mobility domain of the GNEM-FAS instrument a disease-specific measure developed to assess the functional impact of changes in muscle strength on mobility (reflective of the upper extremities). This mobility score ranges from 0 to 40 with higher scores representing greater mobility.
Time Frame: Baseline, Week 48
Population: Primary Analysis Set: participants who had a Baseline and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ace-ER 6 g/Day | Placebo
Number analyzed (Participants) | 45 | 43
units on a scale | -1.40 [-2.21 to -0.58] | -1.08 [-1.86 to -0.29]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day vs Placebo; Test type: Other; p = 0.5608, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.32, 95% CI 2-sided [-1.39 to 0.75] — Difference: Ace-ER 6 g/day - placebo

ADVERSE EVENTS:
Time Frame: Screening through Week 48 plus 28 days (+5 days). The mean (SD) duration of treatment was 340.2 (12.02) days and 332.9 (40.86) days for the Ace-ER and placebo groups, respectively.
Arm/Group | Ace-ER 6 g/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/44
Other Adverse Events (participants affected / at risk) | 38/45 | 30/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=45) | Placebo (N=44)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=45) | Placebo (N=44)
Abdominal distension (Gastrointestinal disorders) | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Flatulence (Gastrointestinal disorders) | 6 | 5
Frequent bowel movements (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 2 | 3
Fatigue (General disorders) | 4 | 4
Influenza like illness (General disorders) | 4 | 11
Pain (General disorders) | 1 | 3
Influenza (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 7
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 7 | 7
Sciatica (Nervous system disorders) | 0 | 3
Sleep disorder (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT02377921/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT02377921/SAP_001.pdf